CLINICAL TRIAL: NCT00788398
Title: Fluid Lavage of Open Wounds (FLOW): A Multi-center, Blinded, Factorial Trial Comparing Alternative Irrigating Solutions and Pressures in Patients With Open Fractures
Brief Title: Fluid Lavage of Open Wounds
Acronym: FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: McMaster University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: GHS-03-08-06; W81XWH-08-1-0473
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Open Fracture Wounds
MeSH Terms: interventions — Saline Solution; Soaps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Saline, gravity flow (Active Comparator)
  Interventions: Procedure: Saline Solution; Procedure: Gravity Flow Irrigation
- Saline, Low Pressure (Active Comparator)
  Interventions: Procedure: Saline Solution; Procedure: Low Pressure Irrigation
- Saline, High Pressure (Active Comparator)
  Interventions: Procedure: Saline Solution; Procedure: High Pressure
- Soap, Gravity Flow (Active Comparator)
  Interventions: Procedure: Soap solution; Procedure: Gravity Flow Irrigation
- Soap, low pressure (Active Comparator)
  Interventions: Procedure: Soap solution; Procedure: Low Pressure Irrigation
- Soap, high pressure (Active Comparator)
  Interventions: Procedure: Soap solution; Procedure: High Pressure

INTERVENTIONS:
Procedure: Saline Solution — Irrigation with Saline
  Arms: Saline, High Pressure; Saline, Low Pressure; Saline, gravity flow
Procedure: Soap solution — Irrigation with Castile Soap Solution (80 ml per 3L bag of saline)
  Arms: Soap, Gravity Flow; Soap, high pressure; Soap, low pressure
Procedure: Gravity Flow Irrigation — Gravity flow irrigation will be standardized across participating centers as 3L bags of normal saline (alone or with soap solution) suspended 6-8 feet above floor level using an I.V. pole. Irrigation tubing (measuring 1/4 - 3/8 inch inner diameter) will be connected to the 3L bag and secured with a stopcock (or compressive device) until ready for use.
  Arms: Saline, gravity flow; Soap, Gravity Flow
Procedure: Low Pressure Irrigation — Irrigation with the Stryker SurgiLav System. At the low pressure setting delivers 5.9 p.s.i. pressure. The high-flow irrigator tip will be held perpendicular to and 5cm above the wound.
  Irrigation with the Zimmer PulsaVac. For low pressure delivery, the shower tip will be used at the low pressure setting which delivers a pressure of 5.8 p.s.i.
  Arms: Saline, Low Pressure; Soap, low pressure
Procedure: High Pressure — Irrigation with the Stryker SurgiLav System. For the high pressure delivery, the multi-orifice tip will be used at the high setting which delivers a pressure of 30 p.s.i.
  Irrigation with the Zimmer PulsaVac System: For the high pressure delivery the shower tip will be used at the high pressure setting which delivers a pressure of 23 p.s.i.
  Arms: Saline, High Pressure; Soap, high pressure

SUMMARY:
Open fracture wounds are a constant challenge to orthopaedic surgeons, with infections a common complication. There is currently little evidence as to which is the most effective way to wash out these wounds. This study is a multi-center, prospective, randomized study. The infection rates will be compared between irrigation using high pressure versus low pressure versus gravity flow, and also saline versus a soap solution as the irrigation solution. The results from this study will help to determine the best method of washing out open fractures wounds. In this study, all open wounds will be washed out using methods commonly used by orthopaedic surgeons

ELIGIBILITY:
Inclusion Criteria:

1. Men or women who are skeletally mature.
2. Fracture of any extremity with complete radiographs.
3. Open fractures (Gustilo-Anderson Types I-IIIB) (Table 2)*.
4. Fracture requiring operative fixation.
5. Provision of informed consent.

Exclusion Criteria:

1. Open fractures with an associated vascular deficit (Gustilo-Anderson Type IIIC).
2. Known allergy to detergents or castile soap ingredients.
3. Previous wound infection or history of osteomyelitis in the injured extremity.
4. Previous fracture with retained hardware in injured extremity that will interfere with new implant fixation.
5. Surgical delay to operative wound management greater than 24 hours from hospital admission.
6. Use of immunosuppressive medication within 6 months.
7. Immunological deficient disease conditions (e.g. HIV).
8. Fracture of the hand (metacarpals and phalanges).
9. Fracture of the toes (phalanges).
10. Likely problems, in the judgment of the investigators, with maintaining follow-up. We will, for example, exclude patients with no fixed address, those who report a plan to move out of town in the next year, or intellectually challenged patients without adequate family support.
11. Previous randomization in this study or a competing study.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2540 (Actual)
Dates: Start 2009-06; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Re-operation within 12 months post initial surgery to treat an infection, manage a wound healing problem, or promote fracture healing. | within 12 months

SECONDARY OUTCOMES:
Patient function and quality of life measured by the Short Form-12 (SF-12) and the EuroQol-5D | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyle J. Jeray, MD, Principal Investigator — Greenville Hospital System; Bradley Petrisor, MD, Principal Investigator — Hamilton Health Sciences Corporation; Mohit Bhandari, MD, Principal Investigator — McMaster University; Gordan Guyatt, M.D., Principal Investigator — McMaster University
Locations (31):
- United States (14):
  - Univeristy of Alabama at Birmingham, Birmingham, Alabama
  - University of California-Irvine, Orange, California
  - University of California- San Francisco, San Francisco, California
  - Wishard Health Services, Indiana University, Indianapolis, Indiana
  - Lahey Clinic, Burlington, Massachusetts
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - St. Louis University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Miami Valley Hospital/Wright State University, Dayton, Ohio
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
- The Alfred, Prahran, Australia
- Canada (14):
  - Royal Columbian Hospital-New Wesminster, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Winnipeg, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario
  - London Health Sciences, London, Ontario
  - Ottawa Hospital- Civic, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Hospital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Hôpital de l'Enfant-Jésus, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
- Sancheti Institute, Prune, India
- Ulleval University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Tornetta P 3rd, Della Rocca GJ, Morshed S, Jones C, Heels-Ansdell D, Sprague S, Petrisor B, Jeray KJ, Del Fabbro G, Bzovsky S, Bhandari M; FLOW Investigators. Risk Factors Associated With Infection in Open Fractures of the Upper and Lower Extremities. J Am Acad Orthop Surg Glob Res Rev. 2020 Dec 8;4(12):e20.00188. doi: 10.5435/JAAOSGlobal-D-20-00188. PMID 33986214
- [Derived] Prada C, Marcano-Fernandez FA, Schemitsch EH, Bzovsky S, Jeray K, Petrisor B, Bhandari M, Sprague S; FLOW Investigators. Timing and Management of Surgical Site Infections in Patients With Open Fracture Wounds: A Fluid Lavage of Open Wounds Cohort Secondary Analysis. J Orthop Trauma. 2021 Mar 1;35(3):128-135. doi: 10.1097/BOT.0000000000001912. PMID 33105456
- [Derived] Busse JW, Heels-Ansdell D, Makosso-Kallyth S, Petrisor B, Jeray K, Tufescu T, Laflamme Y, McKay P, McCabe RE, Le Manach Y, Bhandari M; Fluid Lavage of Open Wounds Investigators. Patient coping and expectations predict recovery after major orthopaedic trauma. Br J Anaesth. 2019 Jan;122(1):51-59. doi: 10.1016/j.bja.2018.06.021. Epub 2018 Aug 6. PMID 30579406
- [Derived] Sprague S, Tornetta P 3rd, Slobogean GP, O'Hara NN, McKay P, Petrisor B, Jeray KJ, Schemitsch EH, Sanders D, Bhandari M; FLOW Investigators. Are large clinical trials in orthopaedic trauma justified? BMC Musculoskelet Disord. 2018 Apr 20;19(1):124. doi: 10.1186/s12891-018-2029-3. PMID 29678204
- [Derived] Shea P, O'Hara NN, Sprague SA, Bhandari M, Petrisor BA, Jeray KJ, Zhan M, Slobogean GP, Pensy RA; Fluid Lavage in Open Wounds Investigators. Wound Surface Area as a Risk Factor for Flap Complications among Patients with Open Fractures. Plast Reconstr Surg. 2018 Jul;142(1):228-236. doi: 10.1097/PRS.0000000000004418. PMID 29608532
- [Derived] FLOW Investigators; Bhandari M, Jeray KJ, Petrisor BA, Devereaux PJ, Heels-Ansdell D, Schemitsch EH, Anglen J, Della Rocca GJ, Jones C, Kreder H, Liew S, McKay P, Papp S, Sancheti P, Sprague S, Stone TB, Sun X, Tanner SL, Tornetta P 3rd, Tufescu T, Walter S, Guyatt GH. A Trial of Wound Irrigation in the Initial Management of Open Fracture Wounds. N Engl J Med. 2015 Dec 31;373(27):2629-41. doi: 10.1056/NEJMoa1508502. Epub 2015 Oct 8. PMID 26448371
- [Derived] Flow Investigators. Fluid lavage of open wounds (FLOW): design and rationale for a large, multicenter collaborative 2 x 3 factorial trial of irrigating pressures and solutions in patients with open fractures. BMC Musculoskelet Disord. 2010 May 6;11:85. doi: 10.1186/1471-2474-11-85. PMID 20459600